CLINICAL TRIAL: NCT02147028
Title: A Randomized Phase II Trial of Hippocampal Sparing Versus Conventional Whole Brain Radiotherapy After Surgical Resection or Radiosurgery in Favourable Prognosis Patients With 1-10 Brain Metastases
Brief Title: Hippocampal Sparing Whole Brain Radiotherapy vs Conventional Whole Brain Radiotherapy in Patients With Brain Metastases
Acronym: HIPPO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other); The Brain Tumour Charity (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL/12/0512; Cancer Research UK (Other Grant/Funding Number: CRUK/13/017)
Record Dates: First submitted 2014-05-21; First posted 2014-05-26 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Brain Metastases
Keywords: whole brain RT; hippocampal sparing; neurocognitive function
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hippocampal sparing whole brain RT (Experimental): 30 Gy in 10 fractions hippocampal sparing whole brain radiotherapy will be administered by Helical Tomotherapy, IMRT, or VMAT
  Interventions: Radiation: Hippocampal sparing whole brain radiotherapy
- Control: Conventional whole brain RT (Active Comparator): 30 Gy in 10 fractions conventional whole brain radiotherapy will be administered
  Interventions: Radiation: Conventional whole brain radiotherapy

INTERVENTIONS:
Radiation: Hippocampal sparing whole brain radiotherapy — 30 Gy in 10 fractions hippocampal sparing whole brain radiotherapy will be administered by Helical Tomotherapy, IMRT, or VMAT
  Arms: Hippocampal sparing whole brain RT
Radiation: Conventional whole brain radiotherapy — 30 Gy in 10 fractions conventional whole brain radiotherapy will be administered
  Arms: Control: Conventional whole brain RT

SUMMARY:
The purpose of this study is to evaluate whether sparing the hippocampi during whole brain radiotherapy following neurosurgery or stereotactic radiosurgery in patients with brain metastases from a systemic tumour helps preserve brain function.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 16 years
* Karnofsky Performance Status (KPS) ≥ 70
* Brain metastases from systemic malignancy which has been histologically confirmed (from the primary or any metastatic site)
* In total, at most 10 distinct brain metastases based on MRI imaging with contrast at any prior time-points
* Each of the brain metastases to have been treated by complete or incomplete surgical excision or by SRS in line with UK SRS commissioning guidelines which in addition for STS treated patients means:

  * Patient selection for SRS by the appropriate MDT(s),
  * No pressure symptoms which would be best relieved by surgery,
  * Life expectancy from extracranial disease greater than 6 months,
  * Gross tumour volume at time of SRS ≤ 20 cc.
* Ability to comply with the following timelines:

  * Randomisation 1 - 4 weeks (+/- 3 days, but only acceptable if accounting for logistical issues) after neurosurgery or last SRS fraction,
  * Start of WBRT or HS-WBRT 4 - 6 weeks (+ 3 days, but only acceptable if accounting for logistical or planning treatment issues) after neurosurgery or last SRS fraction.
* Ability to complete the NCF test battery (including ability to speak English).
* Willing and able to give consent and to comply with treatment and follow up schedule.

Exclusion Criteria:

* Metastases from small cell carcinoma from any site, haematological malignancy, or central nervous system malignancy,
* Leptomeningeal metastases,
* Contraindication to MRI imaging with contrast,
* Prior radiotherapy to the brain (apart from a single course of SRS for brain metastases completed within 1-4 weeks (+/- 3 days) of randomisation and within 4-6 weeks (+3 days) of start of the HIPPO trial treatment),
* Prior neurosurgery for brain metastases (apart from a single operation within 1-4 weeks (+/- 3 days) of randomisation and within 4-6 weeks (+3 days) of start of HIPPO trial treatment), except that one or more earlier operations not immediately preceding HIPPO trial entry will be allowed if:

  * there is no evidence of residual tumour at the resection site on contrast MRI imaging, or
  * residual tumour at the resection site has been treated by SRS immediately prior to entering the HIPPO trial,
* One or more metastases currently or previously within 5 mm of either hippocampus,
* One or more metastases within the brainstem,
* One or more SRS treated metastases in close proximity to critical normal organs, unless the local investigator is satisfied that the dose already received by the critical organ allows for subsequent delivery of the HIPPO protocol radiotherapy doses,
* Disease specific graded prognostic assessment (DS-GPA) score ≤ 1.0 for any of the histologies for which DS-GPA has been defined,
* Past medical history of dementia which is thought to be unrelated to the brain metastases,
* Women of childbearing potential who are known to be pregnant, or are unwilling to use an acceptable method of contraception from the time of informed consent until completion of the course of radiotherapy.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-08-03 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
Total recall assessed using Hopkins Verbal Learning Test-Revised (HVTLR) at 4 months | 4 months after completion of WBRT or HS-WBRT
  A decline in total recall will be assessed as being clinically significant if there is at least a 5 point decrease in total recall score at 4 months, compared to baseline [Jacobson 1991, Brandt 1998]

SECONDARY OUTCOMES:
Neurocognitive function | 2, 4, 6, 12 and 24 months after completion of WBRT or HS-WBRT
  NCF, using a 30-60 min test battery (Memory - HVLT-R, Wechsler Memory Scale (logical memory subtest), Rey figure test, Wechsler digit span; Attention - Test of Everyday Attention (map search subtest), Trail Making Test (Parts A and B); Language - Graded Naming Test); this may be revised in the light of forthcoming recommendations on NCF assessment in brain metastases trials by the RANO (Revised Assessment in Neuro-oncology) working party
Quality of life | 2, 4, 6, 9, 12, 18 and 24 months after completion of WBRT or HS-WBRT
  Quality of life will be assessed using EORTC QLQ C30 and BN20 and EuroQol EQ-5D questionnaires
Length of time functionally independent | 2, 4, 6, 9, 12, 18 and 24 months after completion of WBRT or HS-WBRT
  The duration of functional independence will be assessed as the time for which the Karnofsky Performance Status ≥ 70
Local control of surgery/SRS treated metastases, local and distant intracranial control (treated and new metastases), and disease control within the hippocampal regions | 2, 4, 6, 9, 12, 18 and 24 months after completion of WBRT or HS-WBRT
  Incidence of metastases within the perihippocampal region, local control, and intracranial control will be assessed on the basis of MRI imaging
Overall survival | followed up until 24 months after completion of WBRT or HS-WBRT
  Date of death will be determined from the medical records, or from the GP
Steroid and antiepileptic medication requirements | 2, 4, 6, 9, 12, 18 and 24 months after completion of WBRT or HS-WBRT
  Steroid and antiepileptic medication use will be recorded in patient diaries and assessed at clinic visits
Acute and late side effects of radiotherapy | 2, 4, 6, 9, 12, 18 and 24 months after completion of WBRT or HS-WBRT
  Acute and late side effects of radiotherapy will be assessed using NCI CTCAE scale v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Gillian Whitfield, MA,MB BS,PhD, Study Chair — The Christie NHS Foundation Trust
Locations (7):
- United Kingdom (7):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, Greater London
  - Addenbrooke's Hospital, Cambridge
  - Royal Surrey County Hospital, Guildford
  - Charing Cross Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham University Hospitals, Nottingham
  - Barking, Havering and Redbridge University Hospitals Nhs Trust, Romford